CLINICAL TRIAL: NCT04028102
Title: Optimization of Initial Fluid Challenge by Cardiac and Lung Ultrasound in Patients With Sepsis
Brief Title: Ultrasound Optimization of Initial Fluid Challenge in Sepsis
Acronym: echosepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-034
Record Dates: First submitted 2019-07-17; First posted 2019-07-22 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Sepsis
Keywords: sepsis; treatment; fluid challenge
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Initial sepsis treatment requires fluid challenge. While the Surviving Sepsis Campaign indicates a 30 ml/kg volume, there is concerns on the efficacy and safety of this fixed volume. The aim of this study is to assess the difference between fluid volume determined par cardiac and lung Ultrasound versus the fixed 30 ml/kg.

DETAILED DESCRIPTION:
Initial sepsis treatment requires fluid challenge (FC). While the Surviving Sepsis Campaign (SSC) indicates a fixed 30 ml/kg volume, there is concerns on the efficacy and safety of this volume.

Actually, the required volume is highly dependent of cardiac and pulmonary comorbidities, infection focus localization and intensity. The importance of the initial volume is crucial: if too low, it could not restore the hemodynamic status, if too high, it could induce a lung edema responsible for an increased morbidity and mortality.

Cardiac Ultrasound (US) has demonstrated its efficacy to approach cardiac output by measuring the velocity-time integral (VTI) in the aortic chamber and its variations induced by the FC. While the VTI induced variation by a 500-ml FC in 20 min is above 10%, the patient is still fluid responsiveness and FC has to be continued. Conversely, when the variation is below 10%, FC has to be stopped.

Lung Ultrasound can detect a sub-clinical pulmonary edema before oxygenation degradation by visualization of diffuses B lines. The combination of both techniques is thus able to individualize the actual needed FC volume.

In patients with sepsis as defined by SEPSIS-3 and with hypotension (MAP < 65 mm Hg or lactate > 2 mmol/l), the FC of saline serum is individualized by the US technique. The volume is compared with the fixed 30 ml/kg.

ELIGIBILITY:
Inclusion Criteria:

* patients >18 years old with sepsis as defined by SEPSIS-3 and with hypotension (MAP < 65 mm Hg or lactate > 2 mmol/l)

Exclusion Criteria:

* documented end-of-life
* pregnancy
* B/B initial profile to the first Lung US

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with sepsis and hypotension in the Emergency Department
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
concordance of fluid volume | 3 hours after FC initiation
  number of patients with delta FC volume > 20% between US technique and the theoretical 30 ml/kg

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France